CLINICAL TRIAL: NCT05734937
Title: Ultrasound Evaluation of Gastric Volume in Pediatric Patients Undergoing Adenotonsillectomy Surgery: a Prospective Cohort Study
Brief Title: Ultrasound Evaluation of Gastric Volume in Pediatric Patients Undergoing Adenotonsillectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, Attending Anesthesiologist, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022/985
Record Dates: First submitted 2023-01-20; First posted 2023-02-21 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Gastric Volume; Aspiration; Nausea; Bleeding
MeSH Terms: conditions — Nausea; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gastric assessment of gastric volume (Experimental): ultrasound assessment of gastric volume in Preoperative and postoperative period in right lateral decubitus position in pediatric patients
  Interventions: Other: gastric assessment of gastric volume

INTERVENTIONS:
Other: gastric assessment of gastric volume — ultrasound assessment of gastric volume is going to bel evaluted in the Preoperative and postoperative period while the patients lay in right lateral decubitus position.

SUMMARY:
Adenoidectomy and/or tonsillectomy are performed for many reasons such as recurrent tonsil and adenoid infections, sleep apnea, symptomatic adenotonsillar hypertrophy, halitosis, peritonsillar abscess, and it is one of the most performed surgeries in the world. Passive blood loss from the surgical field into the gastric area may occur during the surgery.

Investigators wonder whether the amount of blood and fluid accumulated in the stomach after tonsillectomy and/or adenoidectomy in children will increase the risk of aspiration. For this purpose, the aim is to compare the results with values considered risky for aspiration by evaluating the pre- and postoperative gastric volume with ultrasound in children who underwent elective adenoidectomy and /or tonsillectomy.

DETAILED DESCRIPTION:
Tonsillectomy and/or adenoidectomy are performed for many reasons such as recurrent tonsil and adenoid infections, sleep apnea, symptomatic adenotonsillar hypertrophy, halitosis, peritonsillar abscess, and it is one of the most performed surgeries in the world. During these operations, there may be fluid and blood accumulation in the stomach.

Investigators wonder whether the amount of blood and fluid accumulated in the stomach after tonsillectomy and/or adenoidectomy in children will increase the risk of aspiration. For this purpose, the aim is to compare the results with values considered risky for aspiration by evaluating the pre- and postoperative gastric volume with ultrasound in children who underwent tonsillectomy and/or adenoidectomy.

This study will include ASA 1,2,3 patients under the age of 18 who will undergo tonsillectomy and/or adenoidectomy in the operating rooms of Istanbul University, Istanbul Medical Faculty, Department of Otorhinolaryngology, after the approval of the ethics committee. All the patients will be given oral midazolam at a dose of 0.3 mg/kg as standard in the preoperative preparation room. After standard monitoring (ECG, NIBP, SpO2) is performed in the operating room, gastric volume will be evaluated by ultrasound in the right lateral position before the operation. After induction of general anesthesia (sevoflurane + 02 + NO2 inhalation, 1 mcg/kg fentanyl, 0.5 mg/kg rocuronium) patients will be intubated. After intubation, gastric volume will be re-evaluated by ultrasound in the right lateral position. anesthesia will be maintained with a mixture of sevoflurane + 40%/60% O2/NO2 for a MAC of 1.0. At the end of the surgery, before the patient is extubated, the gastric volume will be evaluated by ultrasound in the right lateral position. Afterwards, the patients will be extubated and taken to the postoperative recovery room. Nausea and vomiting of patients during awakening and for the next 24 hours will be recorded. Patients' age, gender, height, weight, duration of surgery will also be recorded in the follow-up form.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective adenotonsillectomy surgery overnight fasting
* 1-18 years of age
* Accepting to the join the study
* American Society of Anesthesiology (ASA) classification I-II-III

Exclusion Criteria:

* Age older than 18 years
* Preoperative vomiting or antiemetic medication therapy
* Intubation more than needing more than two laryngoscopy attempts
* Not given approval from the parents
* Disease or conditions affecting gastric volume or motility

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Gastric volume (ml/kg) | During the operation
  Gastric volumes are going to be calculated

SECONDARY OUTCOMES:
The cross sectional area (ACSA) (preoperative)(mm2) | preoperative
  measurements are done with USG and calculated with this formula CSA=(AP(anterior -posterior) diameter x CC(craniotomy-caudal ) diameter x 3.14)/4
The cross sectional area (ACSA) (after intubation)(mm2) | immediately after intubation
  measurements are done with USG and calculated with this formula CSA=(AP(anterior -posterior) diameter x CC(craniotomy-caudal ) diameter x 3.14)/4
The cross sectional area (ACSA) (postoperative)(mm2) | 10 minutes before extubation
  measurements are done with USG and calculated with this formula CSA=(AP(anterior -posterior) diameter x CC(craniotomy-caudal ) diameter x 3.14)/4
postoperative presence and severity of PONV | at the first, second and 24th hours in PACU and at the ward.
  The severity of PONV was assessed according to the four points score :
  None (0 point) nausea (1 point) , nausea with maximum of two vomiting episodes (2 points) , more than two vomiting episodes (3 points)
blood volume in suction system | intraoperative
  weighing sponge, pad, and blood volume in the aspirator
duration of surgery | Intraoperative (throughout the surgical procedure)
  the time from the start of the surgery to the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Öztürk, Resident, Principal Investigator — Istanbul University; Demet Altun, Assoc. Prof, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Desgranges FP, Gagey Riegel AC, Aubergy C, de Queiroz Siqueira M, Chassard D, Bouvet L. Ultrasound assessment of gastric contents in children undergoing elective ear, nose and throat surgery: a prospective cohort study. Anaesthesia. 2017 Nov;72(11):1351-1356. doi: 10.1111/anae.14010. Epub 2017 Aug 14. PMID 28805238
- [Background] Zhang G, Huang X, Shui Y, Luo C, Zhang L. Ultrasound to guide the individual medical decision by evaluating the gastric contents and risk of aspiration: A literature review. Asian J Surg. 2020 Dec;43(12):1142-1148. doi: 10.1016/j.asjsur.2020.02.008. Epub 2020 Mar 11. PMID 32171605
- [Background] Bisinotto FM, Pansani PL, Silveira LA, Naves AA, Peixoto AC, Lima HM, Martins LB. Qualitative and quantitative ultrasound assessment of gastric content. Rev Assoc Med Bras (1992). 2017 Feb;63(2):134-141. doi: 10.1590/1806-9282.63.02.134. PMID 28355374